CLINICAL TRIAL: NCT05627596
Title: Effectiveness of Nicotine Replacement Therapy Sampling in Dental Practices
Brief Title: Free Samples for Health
Acronym: FreSH
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: Medical University of South Carolina (Other); Massachusetts General Hospital (Other); Northwestern University (Other); HealthPartners Institute (Other); University of Alabama at Birmingham (Other); Kaiser Permanente (Other); University of Rochester (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: UH3DE029973 (NIH); UH3DE029973 (NIH)
Record Dates: First submitted 2022-11-16; First posted 2022-11-25 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Electric Toothbrush (Active Comparator): Participants will receive the Ask-Advise-Refer intervention which includes an oral health practitioner asking about their tobacco use, advising them to quit smoking, and referring them to the state quitline. They will also receive a sample bag including information about smoking and oral health, the state quitline, and an electric toothbrush.
  Interventions: Behavioral: Ask-Advise-Refer
- Nicotine Replacement Therapy (Experimental): Participants will receive the Ask-Advise-Refer intervention which includes an oral health practitioner asking about their tobacco use, advising them to quit smoking, and referring them to the state quitline. They will also receive a sample bag including information about smoking and oral health, the state quitline, and a two week supply of 14mg nicotine patches and 4mg lozenges.
  Interventions: Behavioral: Ask-Advise-Refer; Drug: Nicotine Patch, 14 Mg/24 Hr Transdermal Film, Extended Release; Drug: Nicotine lozenge

INTERVENTIONS:
Behavioral: Ask-Advise-Refer — All patients will be asked if they smoke, advised to quit, and referred to the state quitline
Drug: Nicotine Patch, 14 Mg/24 Hr Transdermal Film, Extended Release — 14 mg transdermal nicotine patch
  Arms: Nicotine Replacement Therapy
Drug: Nicotine lozenge — 4mg nicotine lozenge
  Arms: Nicotine Replacement Therapy

SUMMARY:
The Free Samples for Health (FreSH) study tests whether providing free samples of stop smoking medicine called nicotine replacement therapy at dental visits results in a greater number of people quitting smoking than providing a gift of equal value (an electric toothbrush).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* smokes at least 1 combustible cigarette per day on at least 25 days of the month

Exclusion Criteria:

* does not own a smartphone with internet access
* myocardial infarction or stroke in the past 3 months
* pregnant or breastfeeding
* use of tobacco cessation medication in the past week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2025-05-28 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
7-day biochemically confirmed point prevalence abstinence | 6 months post baseline
  Proportion reporting no smoking in the 7 days prior to the 6-month follow-up timepoint and having an exhaled carbon monoxide value of less than 6 parts per million

SECONDARY OUTCOMES:
7-day self-reported point prevalence abstinence | 1 month post baseline
  Proportion reporting no smoking in the 7 days prior to the 1-month follow-up
7-day self-reported point prevalence abstinence | 1 month post baseline
  Proportion reporting no smoking in the 7 days prior to the 3-month follow-up
24-hour intentional quit attempts | 6 months post baseline
  proportion reporting a quit attempt of 24 hours or longer in duration over the course of the study
Smoking heaviness | 6 months post baseline
  Change in cigarettes smoked per day from baseline to the 6 month follow-up
Nicotine replacement therapy utilization | 6 months post baseline
  Proportion reporting using nicotine patch or nicotine lozenge in the 6 months following baseline
Perceived nicotine replacement therapy safety | 6 months post baseline
  Change in self-reported perception of nicotine replacement therapy safety from baseline to 6-month follow-up
Perceived nicotine replacement therapy efficacy | 6 months post baseline
  Change in self-reported perception of nicotine replacement therapy efficacy from baseline to 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Japuntich, Principal Investigator — Hennepin Healthcare/University of Minnesota Medical School
Locations (1):
- Hennepin Healthcare Research Institute, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Fang P, Adkins-Hempel M, Lischka T, Basile S, Rindal DB, Carpenter MJ, Kopycka-Kedzierawski DT, Dahne J, Helseth SA, Levy DE, Truong A, Leo MC, Funkhouser K, Louis DR, Japuntich SJ; National Dental PBRN Collaborative group. A National Dental Practice-Based Research Network phase II, cluster-randomized clinical trial assessing nicotine replacement therapy sampling in dental settings: study protocol for the Free Samples for Health (FreSH) study. BMC Oral Health. 2024 Aug 28;24(1):1007. doi: 10.1186/s12903-024-04758-w. PMID 39198824